CLINICAL TRIAL: NCT07170007
Title: Physiotherapeutic Protocol Compared to Usual Care in the Treatment of Postpartum Primiparas After Perineal Trauma: A Type 1 Hybrid Effectiveness-Implementation Randomized Controlled Trial With Economic Evaluation
Brief Title: Physiotherapeutic Protocol Compared to Usual Care in the Treatment of Primiparas After Perineal Trauma
Acronym: MPR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Caroline Soares de Paula, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10750271
Record Dates: First submitted 2025-08-19; First posted 2025-09-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Episiotomy; Lacerations Perineal; Obstetric Anal Sphincter Injury; Perineal Injury; Perineal Laceration, Tear, or Rupture During Delivery; Perineal Pain; Perineal Tear Resulting From Childbirth; Perineal Tear and Episiotomy
Keywords: pelvic floor dysfunction; woman's health; perineal pain; vaginal birth; perineal tear; postpartum
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, randomized controlled trial with two arms: an intervention group receiving a physiotherapeutic protocol and a control group receiving usual postpartum care. Participants will be randomly allocated, and outcome assessors will be blinded to group assignment. The study follows a Type 1 hybrid effectiveness-implementation design and includes an economic evaluation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in this group will be selected from among primiparous women aged 18 or over, who have suffered a perineal laceration of grade 2 or above or episiotomy, with ≥37 weeks of gestation at the time of delivery, with no history of neurological diseases, and without perineal diseases. According to the 10-group Robson Classification System, only women belonging to group 1 and group 2a will be included. This arm will receive standard postpartum care for perineal trauma from the maternity hospital.
  Interventions: Other: Usual maternity care
- Intervention Group (Experimental): Participants in this group will be selected from among primiparous women aged 18 or over, who have suffered a perineal laceration of grade 2 or above or episiotomy, with ≥37 weeks of gestation at the time of delivery, with no history of neurological diseases, and without perineal diseases. According to the 10-group Robson Classification System, only women belonging to group 1 and group 2a will be included. The women randomized to the Intervention Group the physiotherapeutic protocol (pelvic floor muscle training and cryotherapy, starting in the imediate postpartum and lasting 3 months).
  Interventions: Other: Physiotherapeutic protocol

INTERVENTIONS:
Other: Physiotherapeutic protocol — The women randomized to the Intervention Group will receive the following interventions:
  During hospitalization: Pelvic Floor Muscle Contraction, observing the participant's ability to contract and advising on how to perform it, associated with cryotherapy and information on physiotherapy in women's health, pelvic floor muscles and its dysfunctions, as well as guidance on the care to be taken during hospitalization and after discharge, including guidance on postures to be adopted or avoided, breathing control, load management, intimate hygiene and the use of cryotherapy at home for pain relief.
  After hospitalization, up to 3 months after delivery: Pelvic Floor Muscle Training in weekly online sessions and guidance to carry out the training daily at home, with the same protocols and without supervision. A total of 12 individual online sessions.
  Arms: Intervention Group
Other: Usual maternity care — Participants in the control group will receive standard postpartum care for perineal trauma from the maternity hospital, which includes suturing the injury and oral analgesic medication.
  Arms: Control Group

SUMMARY:
The aim of this study is to assess the effectiveness of a pelvic floor muscle training (PFMT) protocol associated with cryotherapy initiated in the immediate postpartum period in relieving pain in primiparous women who suffered perineal trauma during vaginal delivery. This is a hybrid effectiveness-implementation type 1 randomized controlled trial with economic evaluation, which will include 82 primiparous women who suffered a perineal tear of grade 2 or above or episiotomy during vaginal delivery. The study participants will be selected from among the women who gave birth at the Hospital das Clínicas in Ribeirão Preto and will be randomly assigned to participate in one of two study groups: the Control Group will receive the usual maternity care, that includes suturing the injury and analgesic medication, and the Intervention Group will receive the usual care combined with a physiotherapy protocol of PFMT and cryotherapy, starting in the immediate postpartum period and lasting 3 months. The primary outcome of the study will be the change in perineal pain intensity assessed using an 11-point Numerical Rating Scale; and the secondary outcomes will be self-reported pelvic floor dysfunction, recovery from injury, functionality, health-related quality of life, use of pain medication, genital self-image and implementation outcomes (satisfaction, acceptability, adequacy, feasibility, equity and adherence to the protocol). Assessments will be carried out by a group of health professionals, including physiotherapists and physicians, at 11 points up to 6 months after delivery. Two doctors from the service will be responsible for carrying out the transperineal ultrasound examination to assess the injury, which will be sent to a third international collaborating physician (SD) to assess the results blindly. The other assessments will be carried out by two physiotherapists.Descriptive statistics will be used, including the ANOVA test to confirm homogeneity between the groups, the chi-square test or Fisher's test for categorical variables and Student's t-test or Wilcoxon's non-parametric test for independent samples for quantitative variables.

DETAILED DESCRIPTION:
This study is a type 1 hybrid randomised controlled clinical trial of effectiveness-implementation, with economic evaluation and blinded assessor, which aims to assess the effectiveness and cost-effectiveness of a physiotherapy protocol that combines pelvic floor muscle training (PFMT) with cryotherapy, initiated immediately after vaginal delivery in primiparas who have suffered perineal laceration grade 2 or above or episiotomy.

Eighty-two women who gave birth at the Hospital das Clínicas of the Ribeirão Preto Medical School - USP will be recruited. Participants will be randomised into two groups: Control Group, which will receive only the usual maternity care (analgesic medication and sutures); and Intervention Group, which will receive, in addition to the usual care, the physiotherapy protocol.

The physiotherapy protocol consists of one in-person session during hospitalisation, which will include 20 minutes of cryotherapy and initial instructions on pelvic floor muscle contraction (PFM). After hospital discharge, 12 weekly PFMT sessions will be conducted remotely (online), with guidance for daily continuation of home exercises and application of cryotherapy as needed for perineal pain relief.

The primary outcome will be the intensity of perineal pain, assessed using an 11-point numerical rating scale at the following times: 6-10 hours postpartum, 30 minutes after initial intervention, weekly in the first month, fortnightly in the second month, and at 3 and 6 months postpartum.

Secondary outcome measures include self-reported pelvic floor dysfunction (Australian Pelvic Floor Questionnaire and Wexner Scale), anatomical and functional recovery of the PFM (transperineal ultrasound and vaginal palpation using the modified Oxford scale), functionality (International Physical Activity Questionnaire - IPAQ and functional limitation numerical scale), health-related quality of life (EQ-5D-3L), use of analgesic medications, genital self-image (Female Genital Self-image Scale), gender-based violence (WHO-adapted questionnaire), and implementation outcomes (acceptability, adequacy, feasibility, and adherence to the protocol).

In addition, a comprehensive economic analysis will be conducted from the perspective of society, with a time horizon of 6 months, including cost-effectiveness analysis (clinical outcome: pain intensity) and cost-utility analysis (QALY). The costs evaluated will include interventions, health resources used (medications, tests, medical consultations, and additional physiotherapy sessions), complementary expenses (transportation and caregiver), and loss of productivity.

This protocol may offer a safe, non-pharmacological, effective, and potentially cost-effective intervention for the relief of perineal pain and prevention of pelvic floor dysfunction in primiparous women after vaginal delivery with perineal trauma, and may contribute significantly to public policies and clinical practices in the Brazilian Unified Health System (SUS).

ELIGIBILITY:
Inclusion Criteria:

* The study will include female at birth aged 18 years or older, primiparous (no previous pregnancy after 16 weeks), who have suffered a perineal laceration of grade ≥2 or episiotomy, with ≥37 weeks of gestation at the time of delivery, who have not used testosterone in the last 6 months, with preserved cognitive ability, no history of neurological diseases, no symptoms of vaginal or urinary tract infection and no perineal diseases such as fistulas, genital mutilation, previous perineal surgery for pelvic floor dysfunction or Crohn's disease. According to the Robson 10-Group Classification System, only women belonging to group 1 (nulliparous women with a single vital cephalic pregnancy, ≥37 weeks of gestation in spontaneous labor) and group 2a (nulliparous women with a single vital cephalic pregnancy, ≥37 weeks of gestation who had labor induced) will be included in the study.

Exclusion Criteria:

* Women with conditions such as severe pre-eclampsia or infections, sick newborns or women who refuse to take part in the study will not be included. Participation is voluntary and participants can withdraw from the study at any time.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in perineal pain intensity | Up to 6 months postpartum
  The change in the intensity of perineal pain will be assessed using an 11-point numerical rating scale (NRS), in which the participant will quantify her level of pain on a scale of 0 to 10, where 0 means no pain and 10 means the worst pain imaginable; a change of 2 points in the NRS will be considered clinically significant. The pain assessment will be done by asking the participants: "What is the level of pain in your intimate area at the moment?" and "Do you believe you have taken any measures that could have improved or worsened your pain today?". If the answer is yes, the participant will be asked to specify the measure she believes has worsened or relieved the pain. The assessment will be carried out in person during hospitalization, and after discharge, via text message at the end of the day (around 6pm).

SECONDARY OUTCOMES:
Self-reported symptoms of pelvic floor dysfunction | Up to 6 months postpartum.
  Australian Pelvic Floor Questionnaire, comprising 42 questions in four domains: bladder, bowel, sexual function, and pelvic organ prolapse. The higher the score, the worse the function assessed.
  The bladder section consists of 15 questions, resulting in a final score of 0-45. The bowel section consists of 12 questions, resulting in a final score of 0-34, and the prolapse section consists of 5 questions, resulting in a final score of 0-15, and the sexual function section consists of 10 questions, two qualitative and eight quantitative, with variable scores and a final score of 0-21. A change of 1 point in each section of the scale will be considered clinically significant.
  This assessment will be carried out at four points in time: At baseline; 6-8 weeks after delivery; 3 and 6 months after delivery, remotely.
Anal incontinence | Up to 3 months postpartum.
  The Wexner Scale will be used to assess anal incontinence. The final score ranges from 0 to 20, and the higher the value, the greater the degree of incontinence of the participant. The Wexner scale will be assessed at two points in time: At baseline, and 3 months after delivery.
Integrity of the levator ani muscle | Up to 3 months postpartum
  The integrity of the the levator ani muscle will be assessed using four-dimensional transperineal ultrasound (TPUS). This evaluation is performed offline reconstructing an axial view of the pelvis from the beforementioned ultrasound volume. A tomographic view is used, and the levator ani muscle (LAM) is defined as injured if there is a discontinuity between the LAM and the pubic bone in the plane of minimal hiatal dimension and the 2 slices cranially with 2.5 mm slice intervals. This is evaluated during maximum pelvic floor contraction, or at rest if contraction is not possible. The LAM will be classified as normal, unilateral avulsion, bilateral avulsion. This exam will be performed twice; shortly after birth and 3 months post partum.
Microtrauma of the levator ani muscle | Up to 3 months postpartum
  The integrity of the the levator ani muscle will be assessed using four-dimensional transperineal ultrasound (TPUS). Microtrauma is defined as permanent injury to the muscle fibers without overt avulsion. It is diagnosed during maximum strain (Valsalva maneuver) where a 3D reconstruction of the levator ani muscle (LAM) allows for measuring the levator hiatus (the opening between the puborectalis muscle posterolaterally and the symphysis pubis anteriorly). An area of > 25cm2 is used as a cut off. The results will be presented as total area of the levator hiatus during contraction, relaxation and Valsalva manuever (cm2); anteroposterior diameter of the levator hiatus during contraction, relaxation and Valsalva manuever (mm); transverse diameter of the levator hiatus during contraction, relaxation and Valsalva manuever (mm) This exam will be performed twice; shortly after birth and 3 months post partum.
Obstetric anal sphincter muscle injury (OASI) | Up to 3 months postpartum
  The integrity of the the levator ani muscle will be assessed using four-dimensional transperineal ultrasound (TPUS). The examination intends to evaluate the sphincter apparatus to assess signs of scarring indicating an OASI that has been adequately repaired and of muscle defects indicating either an occult OASI, not identified primarily, or a suboptimal healing.
  These measures are evaluated through the same sonographic method as described above, though an axial plane where 6 slices of equal intervals will be examined. Diagnosis of a persistent sphincter defect is the loss of continuity of the circular internal and/or external sphincter of more than 30 degrees.
  Each slice will be recorded as normal, scar or defect; whenever a defect (>30 degrees) are identified, the size (degrees) are recorded for each of the six slices.
  The presence of a defect in 4 or more of the six slices is defined as an occult OASI. It will be performed shortly after birth and 3 months post partum.
Self-perception | Up to 3 months postpartum
  The self-perception assessment will be carried out using the 'Questionnaire on knowledge and perception of the female pelvic floor', consisting of three parts, which assess the participant's knowledge of the anatomy and function of the pelvic floor muscles, symptoms and treatments for pelvic floor muscle dysfunction, and perception. Each statement has a score ranging from 0 to 3, depending on the statement, generating a maximum score of 40 points. The higher the score obtained, the greater the level of knowledge and perception of contraction and relaxation of the pelvic floor muscles. This assessment will be carried out at baseline and 3 months after delivery.
Function of the pelvic floor muscles | Up to 3 months postpartum
  The assessment of pelvic floor muscle function will also be performed using the Modified Oxford Scale through vaginal palpation. This scale grades pelvic floor muscle function on a scale of 5 degrees, with degree 0: absence of muscle contraction, degree 1: slight muscle contraction; degree 2: weak contraction; degree 3: moderate contraction; degree 4: good contraction; degree 5: strong contraction. Vaginal palpation will be performed with participants in a supine position with knees and hips flexed and abducted and feet resting on the stretcher. Participants will be asked to perform maximum voluntary contraction of the pelvic floor muscles. Participants will be instructed to perform 3 contractions, and the evaluator will rate the last contraction. The higher the score obtained, the better the function of the pelvic floor muscles. This assessment will be carried out after the end of treatment (3 months postpartum), in person.
Functionality | Up to 6 months postpartum.
  Functionality will be assessed by estimating the limitations and restrictions of the parturient in performing activities during hospitalisation and after discharge of participants due to perineal trauma, using a numerical rating scale where 0 represents no difficulty and 10 represents inability to perform the activity; the higher the score, the worse the functionality. The activities questioned will be: turning over in bed, picking up the baby (lying in bed, sitting in bed, standing), breastfeeding (lying down, sitting on the bed, standing), changing the baby, sitting on the bed, getting out of bed, walking, sitting on the toilet, urinating, defecating, performing intimate hygiene after urinating or defecating, getting up from the toilet, and bathing.
  Functionality will be assessed at baseline; 6-8 weeks after delivery; 3 and 6 months after delivery.
Level of physical activity | Up to 6 months postpartum.
  The level of physical activity will be assessed using the International Physical Activity Questionnaire - Short Version, which consists of three questions about daily physical activity, in order to determine the frequency and duration of the activity. The first question relates to strenuous activities (running, playing football, heavy housework), the second to moderate activities (swimming, dancing, gardening). The third question asks how often and for how long the person takes a continuous 10-minute walk.
  Through this questionnaire, participants will be classified as sedentary, insufficiently active, active, or very active.
  This assessment will be carried out at baseline; 6-8 weeks after delivery; 3 and 6 months after delivery.
Health-related quality of life | Up to 6 months postpartum.
  Health-related quality of life will be assessed using the EQ-5D-3L instrument, which comprises two parts: a descriptive system and a visual analog scale. The descriptive system consists of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), where health states are classified with a five-digit number representing the level of severity in each dimension, making it possible to identify 243 health states. The health states identified will be converted into utility using the Brazilian tariff. Utility ranges from -0.2 to 1, with -0.2 representing the worst state of health and 1 representing the best state of health. The visual analog scale ranges from 0 to 100, where participants will self-report their state of health. This assessment will be carried out at baseline; 6-8 weeks after delivery; 3 and 6 months after delivery.
Use of medication | Up to 6 months postpartum.
  Medication use will be monitored in a way that all participants will be asked to record the type and dose of medication used, the duration of intervals and pain before and after administration in a self-reported medication diary that will be provided to participants at baseline, and the blinded evaluator will collect this information via phone calls at the following times: 6-8 weeks after randomization; 3 months after delivery; and 6 months after delivery.
Genital self-image | Up to 3 months postpartum.
  The participants' genital self-image will be assessed using the female genital self-image scale, resulting in a final score that ranges from 7 to 28 points. A score higher than 22 classifies women as satisfied with their genital self-image.
  Genital self-image will be assessed at baseline and 3 months after delivery.
Acceptability | Up to 3 months postpartum
  Acceptability will be assessed using the Intervention Acceptability Measure, which consists of four questions scored from 1 to 5, where 1 means 'strongly disagree' and 5 means 'strongly agree,' resulting in a final score of 4 to 20 points. The higher the score, the better the acceptability. Acceptability will only be assessed 3 months after delivery, or after the last session in the event of dropouts.
Appropriateness | Up to 3 months postpartum
  Appropriateness will be assessed using the Intervention Appropriateness Measure, which consists of four questions scored from 1 to 5, where 1 means 'strongly disagree' and 5 means 'strongly agree,' resulting in a final score of 4 to 20 points. The higher the score, the better the appropriateness. Appropriateness will only be assessed 3 months after delivery, or after the last session in the event of dropouts.
Intervention's feasibility | Up to 3 months postpartum
  Feasibility will be assessed using the Intervention Feasibility Measure, which consists of four questions scored from 1 to 5, where 1 means 'strongly disagree' and 5 means 'strongly agree,' resulting in a final score of 4 to 20 points. The higher the score, the better the feasibility. Feasibility will only be assessed 3 months after delivery, or after the last session in the event of dropouts.
Participant's satisfaction | Up to 3 months postpartum
  The participant's satisfaction with the protocol and its outcome will be assessed using a numerical rating scale scored from 0 to 3, where 0 represents complete dissatisfaction, 1 represents moderate dissatisfaction, 2 represents moderate satisfaction, and 3 represents complete satisfaction, resulting in a final score of 0-15. The higher the score obtained, the greater the satisfaction. Satisfaction will only be assessed 3 months after delivery, or after the last session in the event of dropouts.
Participant's adherence | Up to 3 months postpartum
  The participant's adherence to treatment will be assessed using a questionnaire with questions about the continuous use of resources, participation in online sessions, and the practice of pelvic floor muscle training at home, whether there are any modifications that the participant believes are necessary to the protocol, as well as the retention and dropout rates of participants. In cases of withdrawal, a question about the reason for withdrawal will be added. Adherence will only be assessed 3 months after delivery, or after the last session in the event of dropouts.
Gender-based violence | Up to 3 months postpartum
  Gender-based violence will be assessed using the "Adapted Questionnaire: Multi-Country Study on Women's Health and Domestic Violence (WHO)", composed of 14 questions covering psychological, physical and sexual violence. The assessment of violence will be carried out at baseline and 3 months after delivery, where the latter will include the question "Were you forced to have sexual intercourse before the end of the 40-day protection period?" If the answer is positive, it will be considered sexual violence.
Economic evaluation | Up to 6 months postpartum
  The economic evaluation will be carried out from society's perspective. The costs to society will be made up of the costs of the interventions, health care costs (use of resources consumed by the women), patient/family costs (complementary expenses, informal care and transport costs) and lost productivity (estimated from the hours of absenteeism from work, paid and unpaid, of the woman and her companion), and will be identified by a self-reported cost diary, collected 6 to 8 weeks after randomization, 3 and 6 months after delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results of this study (after de-identification) will be made available upon reasonable request. Data will include variables related to the primary and secondary outcomes, as well as the study protocol and statistical analysis plan. Requests will be evaluated on a case-by-case basis to assess the scientific merit and credibility of the proposal. Access will be granted only to qualified researchers with appropriate ethical approvals and data protection measures in place. Requests should be submitted to the principal investigator at carolinesoarespaula@gmail.com.

REFERENCES:
- [Background] Frawley HC, Galea MP, Phillips BA, Sherburn M, Bo K. Reliability of pelvic floor muscle strength assessment using different test positions and tools. Neurourol Urodyn. 2006;25(3):236-242. doi: 10.1002/nau.20201. PMID 16299815
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Schraiber LB, Latorre Mdo R, Franca I Jr, Segri NJ, D'Oliveira AF. Validity of the WHO VAW study instrument for estimating gender-based violence against women. Rev Saude Publica. 2010 Aug;44(4):658-66. doi: 10.1590/s0034-89102010000400009. English, Portuguese. PMID 20676557
- [Background] Fioratti I, Santos VS, Fernandes LG, Rodrigues KA, Soares RJ, Saragiotto BT. Translation, cross-cultural adaptation and measurement properties of three implementation measures into Brazilian-Portuguese. Arch Physiother. 2023 Mar 27;13(1):7. doi: 10.1186/s40945-023-00160-x. PMID 36967380
- [Background] Arruda, G. T. D., Silva, E. V. D., Somavilla, P., Oliveira, M. C. R. D., & Braz, M. M. (2023). Female Genital Self-image Scale (FGSIS): cut-off point, reliability, and validation of measurement properties in Brazilian women. Fisioterapia e Pesquisa, 30, e22015823en.
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Lu YY, Su ML, Gau ML, Lin KC, Au HK. The efficacy of cold-gel packing for relieving episiotomy pain - a quasi-randomised control trial. Contemp Nurse. 2015;50(1):26-35. doi: 10.1080/10376178.2015.1010257. Epub 2015 Jun 10. PMID 26058405
- [Background] Brennen R, Frawley HC, Martin J, Haines TP. Group-based pelvic floor muscle training for all women during pregnancy is more cost-effective than postnatal training for women with urinary incontinence: cost-effectiveness analysis of a systematic review. J Physiother. 2021 Apr;67(2):105-114. doi: 10.1016/j.jphys.2021.03.001. Epub 2021 Mar 23. PMID 33771484
- [Background] Cacciari LP, Kouakou CR, Poder TG, Vale L, Morin M, Mayrand MH, Tousignant M, Dumoulin C. Group-based pelvic floor muscle training is a more cost-effective approach to treat urinary incontinence in older women: economic analysis of a randomised trial. J Physiother. 2022 Jul;68(3):191-196. doi: 10.1016/j.jphys.2022.06.001. Epub 2022 Jun 23. PMID 35753969
- [Background] Beleza ACS, Ferreira CHJ, Driusso P, Dos Santos CB, Nakano AMS. Effect of cryotherapy on relief of perineal pain after vaginal childbirth with episiotomy: a randomized and controlled clinical trial. Physiotherapy. 2017 Dec;103(4):453-458. doi: 10.1016/j.physio.2016.03.003. Epub 2016 Nov 9. PMID 27956033
- [Background] van der Roer N, Boos N, van Tulder MW. Economic evaluations: a new avenue of outcome assessment in spinal disorders. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S109-17. doi: 10.1007/s00586-005-1052-x. Epub 2005 Dec 1. PMID 16320029
- [Background] Laranjeira FO, Petramale CA. A avaliação econômica em saúde na tomada de decisão: a experiência da CONITEC. BIS, Bol Inst Saúde. 2013;14(2):165-170.
- [Background] Black WC. The CE plane: a graphic representation of cost-effectiveness. Med Decis Making. 1990 Jul-Sep;10(3):212-4. doi: 10.1177/0272989X9001000308. PMID 2115096
- [Background] Willan AR, Briggs AH, Hoch JS. Regression methods for covariate adjustment and subgroup analysis for non-censored cost-effectiveness data. Health Econ. 2004 May;13(5):461-75. doi: 10.1002/hec.843. PMID 15127426
- [Background] Sterne JA, White IR, Carlin JB, Spratt M, Royston P, Kenward MG, Wood AM, Carpenter JR. Multiple imputation for missing data in epidemiological and clinical research: potential and pitfalls. BMJ. 2009 Jun 29;338:b2393. doi: 10.1136/bmj.b2393. PMID 19564179
- [Background] Ben AJ, van Dongen JM, El Alili M, Esser JL, Broulikova HM, Bosmans JE. Conducting Trial-Based Economic Evaluations Using R: A Tutorial. Pharmacoeconomics. 2023 Nov;41(11):1403-1413. doi: 10.1007/s40273-023-01301-7. Epub 2023 Jul 17. PMID 37458913
- [Background] Miyamoto GC, Ben AJ, Bosmans JE, van Tulder MW, Lin CC, Cabral CMN, van Dongen JM. Interpretation of trial-based economic evaluations of musculoskeletal physical therapy interventions. Braz J Phys Ther. 2021 Sep-Oct;25(5):514-529. doi: 10.1016/j.bjpt.2021.06.011. Epub 2021 Jul 21. PMID 34340933
- [Background] MATSUDO S., et al. Questionário internacional de atividade física (IPAQ): Estudo de validade e reprodutibilidade no Brasil. 2001.
- [Background] Menezes Rde M, Andrade MV, Noronha KV, Kind P. EQ-5D-3L as a health measure of Brazilian adult population. Qual Life Res. 2015 Nov;24(11):2761-76. doi: 10.1007/s11136-015-0994-7. Epub 2015 Apr 21. PMID 25896666
- [Background] Bergendahl S, Jonsson M, Hesselman S, Ankarcrona V, Leijonhufvud A, Wihlback AC, Wallstrom T, Rydstrom E, Friberg H, Kopp Kallner H, Brismar Wendel S. Lateral episiotomy or no episiotomy in vacuum assisted delivery in nulliparous women (EVA): multicentre, open label, randomised controlled trial. BMJ. 2024 Jun 17;385:e079014. doi: 10.1136/bmj-2023-079014. PMID 38886011
- [Background] Robson M, Murphy M, Byrne F. Quality assurance: The 10-Group Classification System (Robson classification), induction of labor, and cesarean delivery. Int J Gynaecol Obstet. 2015 Oct;131 Suppl 1:S23-7. doi: 10.1016/j.ijgo.2015.04.026. PMID 26433499
- [Background] Baessler K, Mowat A, Maher CF. The minimal important difference of the Australian Pelvic Floor Questionnaire. Int Urogynecol J. 2019 Jan;30(1):115-122. doi: 10.1007/s00192-018-3724-1. Epub 2018 Aug 7. PMID 30088031
- [Background] Amorim AC, Roque LC, Sartori MGF; GPAP Study Group. Australian Pelvic Floor Questionnaire: translation, cultural adaptation, and validation. Int Urogynecol J. 2023 May;34(5):1001-1006. doi: 10.1007/s00192-022-05447-4. Epub 2023 Jan 27. PMID 36705730
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] Zakariaee SS, Shahoei R, Hashemi Nosab L, Moradi G, Farshbaf M. The Effects of Transcutaneous Electrical Nerve Stimulation on Post-Episiotomy Pain Severity in Primiparous Women: A Randomized, Controlled, Placebo Clinical Trial. Galen Med J. 2019 Aug 14;8:e1404. doi: 10.31661/gmj.v8i0.1404. eCollection 2019. PMID 34466506
- [Background] Polden, M. and J. Mantle, Physiotherapy in obstetrics and gynaecology. (No Title), 1990.
- [Background] de Souza Bosco Paiva C, Junqueira Vasconcellos de Oliveira SM, Amorim Francisco A, da Silva RL, de Paula Batista Mendes E, Steen M. Length of perineal pain relief after ice pack application: A quasi-experimental study. Women Birth. 2016 Apr;29(2):117-22. doi: 10.1016/j.wombi.2015.09.002. Epub 2015 Sep 26. PMID 26395154
- [Background] East CE, Dorward ED, Whale RE, Liu J. Local cooling for relieving pain from perineal trauma sustained during childbirth. Cochrane Database Syst Rev. 2020 Oct 9;10(10):CD006304. doi: 10.1002/14651858.CD006304.pub4. PMID 33034900
- [Background] Neels H, De Wachter S, Wyndaele JJ, Wyndaele M, Vermandel A. Does pelvic floor muscle contraction early after delivery cause perineal pain in postpartum women? Eur J Obstet Gynecol Reprod Biol. 2017 Jan;208:1-5. doi: 10.1016/j.ejogrb.2016.11.009. Epub 2016 Nov 11. PMID 27875777
- [Background] Leeman L, Fullilove AM, Borders N, Manocchio R, Albers LL, Rogers RG. Postpartum perineal pain in a low episiotomy setting: association with severity of genital trauma, labor care, and birth variables. Birth. 2009 Dec;36(4):283-8. doi: 10.1111/j.1523-536X.2009.00355.x. PMID 20002420
- [Background] Cooklin AR, Amir LH, Jarman J, Cullinane M, Donath SM; CASTLE Study Team. Maternal Physical Health Symptoms in the First 8 Weeks Postpartum Among Primiparous Australian Women. Birth. 2015 Sep;42(3):254-60. doi: 10.1111/birt.12168. Epub 2015 Jun 19. PMID 26088503
- [Background] East CE, Sherburn M, Nagle C, Said J, Forster D. Perineal pain following childbirth: prevalence, effects on postnatal recovery and analgesia usage. Midwifery. 2012 Feb;28(1):93-7. doi: 10.1016/j.midw.2010.11.009. Epub 2011 Jan 13. PMID 21236531
- [Background] Lowenstein L, Gruenwald I, Gartman I, Vardi Y. Can stronger pelvic muscle floor improve sexual function? Int Urogynecol J. 2010 May;21(5):553-6. doi: 10.1007/s00192-009-1077-5. Epub 2010 Jan 20. PMID 20087572
- [Background] Braekken IH, Majida M, Ellstrom Engh M, Bo K. Can pelvic floor muscle training improve sexual function in women with pelvic organ prolapse? A randomized controlled trial. J Sex Med. 2015 Feb;12(2):470-80. doi: 10.1111/jsm.12746. Epub 2014 Nov 17. PMID 25401779
- [Background] Gommesen D, Nohr E, Qvist N, Rasch V. Obstetric perineal tears, sexual function and dyspareunia among primiparous women 12 months postpartum: a prospective cohort study. BMJ Open. 2019 Dec 16;9(12):e032368. doi: 10.1136/bmjopen-2019-032368. PMID 31848167
- [Background] Mathe M, Valancogne G, Atallah A, Sciard C, Doret M, Gaucherand P, Beaufils E. Early pelvic floor muscle training after obstetrical anal sphincter injuries for the reduction of anal incontinence. Eur J Obstet Gynecol Reprod Biol. 2016 Apr;199:201-6. doi: 10.1016/j.ejogrb.2016.01.025. Epub 2016 Feb 26. PMID 26963793
- [Background] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Background] Morkved S, Bo K. Effect of pelvic floor muscle training during pregnancy and after childbirth on prevention and treatment of urinary incontinence: a systematic review. Br J Sports Med. 2014 Feb;48(4):299-310. doi: 10.1136/bjsports-2012-091758. Epub 2013 Jan 30. PMID 23365417
- [Background] Kahyaoglu Sut H, Balkanli Kaplan P. Effect of pelvic floor muscle exercise on pelvic floor muscle activity and voiding functions during pregnancy and the postpartum period. Neurourol Urodyn. 2016 Mar;35(3):417-22. doi: 10.1002/nau.22728. Epub 2015 Feb 3. PMID 25648223
- [Background] Du Y, Xu L, Ding L, Wang Y, Wang Z. The effect of antenatal pelvic floor muscle training on labor and delivery outcomes: a systematic review with meta-analysis. Int Urogynecol J. 2015 Oct;26(10):1415-27. doi: 10.1007/s00192-015-2654-4. Epub 2015 Feb 25. PMID 25711728
- [Background] Gomes Lopes L, Maia Dutra Balsells M, Teixeira Moreira Vasconcelos C, Leite de Araujo T, Teixeira Lima FE, de Souza Aquino P. Can pelvic floor muscle training prevent perineal laceration? A systematic review and meta-analysis. Int J Gynaecol Obstet. 2022 May;157(2):248-254. doi: 10.1002/ijgo.13826. Epub 2021 Aug 4. PMID 34270799
- [Background] Dieb AS, Shoab AY, Nabil H, Gabr A, Abdallah AA, Shaban MM, Attia AH. Perineal massage and training reduce perineal trauma in pregnant women older than 35 years: a randomized controlled trial. Int Urogynecol J. 2020 Mar;31(3):613-619. doi: 10.1007/s00192-019-03937-6. Epub 2019 Apr 2. PMID 30941442
- [Background] Jiang H, Qian X, Carroli G, Garner P. Selective versus routine use of episiotomy for vaginal birth. Cochrane Database Syst Rev. 2017 Feb 8;2(2):CD000081. doi: 10.1002/14651858.CD000081.pub3. PMID 28176333
- [Background] Dai S, Chen H, Luo T. Prevalence and factors of urinary incontinence among postpartum: systematic review and meta-analysis. BMC Pregnancy Childbirth. 2023 Oct 28;23(1):761. doi: 10.1186/s12884-023-06059-6. PMID 37898733
- [Background] Mikolajczyk RT, Zhang J, Troendle J, Chan L. Risk factors for birth canal lacerations in primiparous women. Am J Perinatol. 2008 May;25(5):259-64. doi: 10.1055/s-2008-1075040. PMID 18509884
- [Background] Shmueli A, Gabbay Benziv R, Hiersch L, Ashwal E, Aviram R, Yogev Y, Aviram A. Episiotomy - risk factors and outcomes. J Matern Fetal Neonatal Med. 2017 Feb;30(3):251-256. doi: 10.3109/14767058.2016.1169527. Epub 2016 Apr 19. PMID 27018243
- [Background] Vale de Castro Monteiro M, Pereira GM, Aguiar RA, Azevedo RL, Correia-Junior MD, Reis ZS. Risk factors for severe obstetric perineal lacerations. Int Urogynecol J. 2016 Jan;27(1):61-7. doi: 10.1007/s00192-015-2795-5. Epub 2015 Jul 30. PMID 26224381
- [Background] Verghese TS, Champaneria R, Kapoor DS, Latthe PM. Obstetric anal sphincter injuries after episiotomy: systematic review and meta-analysis. Int Urogynecol J. 2016 Oct;27(10):1459-67. doi: 10.1007/s00192-016-2956-1. Epub 2016 Feb 19. PMID 26894605
- [Background] Carroli G, Mignini L. Episiotomy for vaginal birth. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD000081. doi: 10.1002/14651858.CD000081.pub2. PMID 19160176
- [Background] Arnold, K.C., et al., Prevention and management of obstetric lacerations at vaginal delivery. Obstetrics Essentials: A Question-Based Review, 2017: p. 253-259.
- [Background] Abedzadeh-Kalahroudi M, Talebian A, Sadat Z, Mesdaghinia E. Perineal trauma: incidence and its risk factors. J Obstet Gynaecol. 2019 Feb;39(2):206-211. doi: 10.1080/01443615.2018.1476473. Epub 2018 Sep 6. PMID 30187786
- [Background] Smith LA, Price N, Simonite V, Burns EE. Incidence of and risk factors for perineal trauma: a prospective observational study. BMC Pregnancy Childbirth. 2013 Mar 7;13:59. doi: 10.1186/1471-2393-13-59. PMID 23497085
- [Background] Dias BAS, Leal MDC, Esteves-Pereira AP, Nakamura-Pereira M. Variations in cesarean and repeated cesarean section rates in Brazil according to gestational age at birth and type of hospital. Cad Saude Publica. 2022 Jul 15;38(6):e00073621. doi: 10.1590/0102-311XPT073621. eCollection 2022. English, Portuguese. PMID 35857919
- [Background] Rebelo F, da Rocha CM, Cortes TR, Dutra CL, Kac G. High cesarean prevalence in a national population-based study in Brazil: the role of private practice. Acta Obstet Gynecol Scand. 2010 Jul;89(7):903-8. doi: 10.3109/00016349.2010.484044. PMID 20583936
- [Background] Osterman MJK, Hamilton BE, Martin JA, Driscoll AK, Valenzuela CP. Births: Final Data for 2021. Natl Vital Stat Rep. 2023 Jan;72(1):1-53. PMID 36723449
- [Background] Betran AP, Torloni MR, Zhang J, Ye J, Mikolajczyk R, Deneux-Tharaux C, Oladapo OT, Souza JP, Tuncalp O, Vogel JP, Gulmezoglu AM. What is the optimal rate of caesarean section at population level? A systematic review of ecologic studies. Reprod Health. 2015 Jun 21;12:57. doi: 10.1186/s12978-015-0043-6. PMID 26093498
- [Background] Chen C, Yan Y, Gao X, Xiang S, He Q, Zeng G, Liu S, Sha T, Li L. Influences of Cesarean Delivery on Breastfeeding Practices and Duration: A Prospective Cohort Study. J Hum Lact. 2018 Aug;34(3):526-534. doi: 10.1177/0890334417741434. Epub 2018 Jan 24. PMID 29365288
- [Background] Sandall J, Tribe RM, Avery L, Mola G, Visser GH, Homer CS, Gibbons D, Kelly NM, Kennedy HP, Kidanto H, Taylor P, Temmerman M. Short-term and long-term effects of caesarean section on the health of women and children. Lancet. 2018 Oct 13;392(10155):1349-1357. doi: 10.1016/S0140-6736(18)31930-5. PMID 30322585
- [Background] Mascarello KC, Horta BL, Silveira MF. Maternal complications and cesarean section without indication: systematic review and meta-analysis. Rev Saude Publica. 2017;51:105. doi: 10.11606/S1518-8787.2017051000389. Epub 2017 Nov 17. PMID 29166440
- [Background] Sharma S, Dhakal I. Cesarean vs Vaginal Delivery : An Institutional Experience. JNMA J Nepal Med Assoc. 2018 Jan-Feb;56(209):535-539. PMID 30058639
- [Background] Juliato CRT. Impact of Vaginal Delivery on Pelvic Floor. Rev Bras Ginecol Obstet. 2020 Feb;42(2):65-66. doi: 10.1055/s-0040-1709184. Epub 2020 Mar 30. No abstract available. PMID 32227320
- [Background] Gregory KD, Jackson S, Korst L, Fridman M. Cesarean versus vaginal delivery: whose risks? Whose benefits? Am J Perinatol. 2012 Jan;29(1):7-18. doi: 10.1055/s-0031-1285829. Epub 2011 Aug 10. PMID 21833896
- [Background] Handa VL, Blomquist JL, Knoepp LR, Hoskey KA, McDermott KC, Munoz A. Pelvic floor disorders 5-10 years after vaginal or cesarean childbirth. Obstet Gynecol. 2011 Oct;118(4):777-84. doi: 10.1097/AOG.0b013e3182267f2f. PMID 21897313
- [Background] Moossdorff-Steinhauser HFA, Berghmans BCM, Spaanderman MEA, Bols EMJ. Prevalence, incidence and bothersomeness of urinary incontinence in pregnancy: a systematic review and meta-analysis. Int Urogynecol J. 2021 Jul;32(7):1633-1652. doi: 10.1007/s00192-020-04636-3. Epub 2021 Jan 13. PMID 33439277
- [Background] Bozkurt M, Yumru AE, Sahin L. Pelvic floor dysfunction, and effects of pregnancy and mode of delivery on pelvic floor. Taiwan J Obstet Gynecol. 2014 Dec;53(4):452-8. doi: 10.1016/j.tjog.2014.08.001. PMID 25510682
- [Background] National Guideline Alliance (UK). Assessment in non-specialist care: Pelvic floor dysfunction: prevention and non-surgical management: Evidence review I. London: National Institute for Health and Care Excellence (NICE); 2021 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK579555/ PMID 35438877
- [Background] DeLancey JO. The hidden epidemic of pelvic floor dysfunction: achievable goals for improved prevention and treatment. Am J Obstet Gynecol. 2005 May;192(5):1488-95. doi: 10.1016/j.ajog.2005.02.028. PMID 15902147
- [Background] Eickmeyer SM. Anatomy and Physiology of the Pelvic Floor. Phys Med Rehabil Clin N Am. 2017 Aug;28(3):455-460. doi: 10.1016/j.pmr.2017.03.003. Epub 2017 May 27. PMID 28676358
- See also: Related Info — https://www.ibge.gov.br/
- See also: Related Info — http://sigtap.datasus.gov.br/tabela-unificada/app/sec/inicio.jsp

DOCUMENTS (3):
  • Study Protocol (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT07170007/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT07170007/SAP_001.pdf
  • Informed Consent Form (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT07170007/ICF_002.pdf